CLINICAL TRIAL: NCT00606489
Title: A Multicenter, Randomized, Double-blind, Placebo-Controlled Trial of Ibuprofen Injection (IVIb) for Treatment of Fever and Pain in Burn Patients
Brief Title: Efficacy and Safety Study of Caldolor (Intravenous Ibuprofen) in Hospitalized Adult and Pediatric Burn Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cumberland Pharmaceuticals (Industry)
Responsible Party: Amy Rock, Ph.D., Senior Manager, Regulatory Affairs, Cumberland Pharmaceuticals Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CPI-CL-010
Record Dates: First submitted 2008-01-22; First posted 2008-02-04 (Estimated); Results first posted 2011-08-11 (Estimated); Last update posted 2011-08-11 (Estimated); Status verified 2011-07

CONDITIONS: Burns
MeSH Terms: conditions — Burns | interventions — Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Placebo Comparator)
  Interventions: Drug: Placebo
- 2 (Experimental)
  Interventions: Drug: Caldolor

INTERVENTIONS:
Drug: Caldolor — 800 milligrams of intravenous ibuprofen (patients greater 12 years of age) or 10 milligrams/kilograms (patients greater than 12 years; maximum of 400 milligrams) every 6 hours
  Arms: 2
Drug: Placebo — Placebo
  Arms: 1

SUMMARY:
The primary objective of this study of Caldolor administered to hospitalized adult and pediatric burn patients is to determine the efficacy of Caldolor on reducing fever when compared to placebo when administered every 6 hours for at least 24 hours.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with second and/or third degree thermal burns covering more than 10 percent total body surface area (including face) with anticipated hospital stay greater than 72 hours.
2. Adequate intravenous access
3. Have fever, documented by temperature greater than or equal to 38.0 degree celsius (100.4 degree fahrenheit)

Exclusion Criteria:

1. Patients with electric burns
2. Use of acetaminophen, non-steriodal anti-inflammatory agents (NSAIDs) or other fever reducing medications within 4 hours prior to dosing
3. Patients taking warfarin or lithium
4. Active, clinically significant asthma
5. History of allergy or hypersensitivity to any component of intravenous ibuprofen, NSAIDs, aspirin (or related products), or COX-2 inhibitors
6. Pregnant or nursing
7. History of severe head trauma that required current hospitalization, intracranial surgery or stroke within the previous 30 days, or any history of intracerebral arteriovenous malformation, cerebral aneurism or central nervous system mass lesion
8. Have a history of congenital bleeding diathesis (e.g. hemophilia) or any active clinically significant bleeding, or have underlying platelet dysfunction including (but not limited to) idiopathic thrombocytopenic purpura, disseminated intravascular coagulation, or congenital platelet dysfunction
9. Have gastrointestional bleeding that required medical intervention within the previous 6 weeks (unless definitive surgery has been performed)
10. Have a platelet count less than 20,000 mm^3
11. Be on dialysis
12. Be receiving full dose anticoagulation therapy or Activated Protein C within 6 hours before dosing (clopidogrel, prophylaxis with enoxaparin or subcutaneous heparin is acceptable)
13. Inability to understand the requirements of the study, be willing to provide written informed consent (as evidenced by signature on an informed consent document approved by an Institutional Review Board [IRB]), and agree to abide by the study restrictions (If the patient is incapacitated, informed consent will be sought from a legally acceptable representative.)
14. Refusal to provide written authorization for use and disclosure of protected health information (If the patient is incapacitated, informed consent will be sought from a legally acceptable representative.)
15. Have received another investigational drug within the past 30 days
16. Be otherwise unsuitable for the study in the opinion of the investigator

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2007-11; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (2):
  - Orlando Regional Medical Center, Orlando, Florida
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
- India (3):
  - Naik's Hospital, Baroda, Kothi
  - Lokmanya Tilak Municipal Medical College, Mumbai, Sion
  - Surya Hospitals Pvt. Ltd, Pune

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were patients admitted to the study centers who had second and third degree thermal burns covering more than 10% total body surface area, including the face.
Period: Overall Study
Arm/Group | Placebo (250 Milliliters Normal Saline) | 800mg Intravenous Ibuprofen
Started | 21 | 40
Completed | 21 | 40
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo (250 Milliliters Normal Saline) | 800mg Intravenous Ibuprofen | Total
Number analyzed (Participants) | 21 | 40 | 61
Age Continuous [Mean (Standard Deviation); unit: years] | 30 (11.9) | 33 (10.8) | 32 (11.2)
Age, Customized [Number; unit: participants]
  <=12 years old | 0 | 0 | 0
  >12 years old | 21 | 40 | 61
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 25 | 36
  Male | 10 | 15 | 25
Region of Enrollment [Number; unit: participants]
  United States | 7 | 9 | 16
  India | 14 | 31 | 45

OUTCOME MEASURES:

1. Primary Outcome: Temperature
Description: Area under the curve temperature from baseline to hour 24 following initiation of treatment.
Time Frame: 0 to 24 hours
Population: Efficacy analyses were performed on the Intent to Treat (ITT) population and the Efficacy Evaluable Population (EEP). All randomized patients who received at least a partial dose of CTM were included in the ITT analyses. All data below represents the ITT analyses.
Measure: Least Squares Mean (Standard Error); unit: Degree Celcius times hours (AUC-T)
Arm/Group | Placebo (250 Milliliters Normal Saline) | 800mg Intravenous Ibuprofen
Number analyzed (Participants) | 21 | 40
Degree Celcius times hours (AUC-T) | 18.29 (2.2) | 12.21 (1.7)

ADVERSE EVENTS:
Arm/Group | Placebo (250 Milliliters Normal Saline) | 800mg Intravenous Ibuprofen
Serious Adverse Events (participants affected / at risk) | 3/21 | 5/40
Other Adverse Events (participants affected / at risk) | 15/21 | 23/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (250 Milliliters Normal Saline) (N=21) | 800mg Intravenous Ibuprofen (N=40)
Cardiopulmonary arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Acute respiratory arrest syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Severe septic shock (Infections and infestations) | 0 (0) | 1 (1)
Invasive wound sepsis (Infections and infestations) | 0 (0) | 1 (1)
Breathlessness (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Septicemia (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (250 Milliliters Normal Saline) (N=21) | 800mg Intravenous Ibuprofen (N=40)
Leukocytosis (Blood and lymphatic system disorders) | 4 (4) | 6 (6)
Anemia (Blood and lymphatic system disorders) | 3 (3) | 5 (5)
Hyperchloremia (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Hypotension (Vascular disorders) | 2 (2) | 5 (5)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Cellulitis (Infections and infestations) | 2 (2) | 1 (1)
Hyperthermia (General disorders) | 1 (1) | 2 (2)
Hyperpyrexia (General disorders) | 2 (2) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1)
Acute respiratory distress syndrom (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No